CLINICAL TRIAL: NCT05037097
Title: A Phase 1/2 Randomized, Observer-Blind Study of the Safety, Reactogenicity, and Immunogenicity of 3 SARS-CoV-2 RNA Vaccine Candidates in Adults Previously Vaccinated and Not Previously Vaccinated Against SARS-CoV-2
Brief Title: A Trial Evaluating the Safety and Immunogenicity of 3 COVID-19 SARS-CoV-2 RNA Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARCT-165-01
Record Dates: First submitted 2021-08-30; First posted 2021-09-08 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; SARS-CoV-2 Infection; Corona Virus Infection
Keywords: SARS-CoV-2 Vaccine; Coronavirus Virus Diseases; RNA COVID-19; COVID-19 Vaccine Arcturus; Self Amplifying RNA Vaccine; Variants of Concern
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — ARCT-154 vaccine

STUDY DESIGN:
Intervention Model Description: The study will evaluate 3 investigational vaccines in parallel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Study Group 1, Adult Participants Seronegative, Not Previously Vaccinated randomized to ARCT-165 (Experimental): Participants will receive one dose of ARCT-165 on Day 1 and one dose of ARCT-165 on Day 29
  Interventions: Biological: ARCT-165
- Study Group 2, Adult Participants Seronegative, Not Previously Vaccinated randomized to ARCT-154 (Experimental): Participants will receive one dose of ARCT-154 on Day 1 and one dose of ARCT-154 on Day 29
  Interventions: Biological: ARCT-154
- Study Group 3, Adult Participants Seronegative, Not Previously Vaccinated to receive ARCT-021 (Experimental): Participants will receive one dose of ARCT-021 on Day 1 and one dose of ARCT-021 on Day 29
  Interventions: Biological: ARCT-021
- Study Group 4, Adult Participants Seropositive, Not Previously Vaccinated to receive ARCT-021 (Experimental): Participants will receive one dose of ARCT-021 on Day 1 and one dose of ARCT-021 on Day 29
  Interventions: Biological: ARCT-021
- Study Group 5, Adult Participants Seropositive, Not Previously Vaccinated randomized to ARCT-154 (Experimental): Participants will receive one dose of ARCT-154 on Day 1 and one dose of ARCT-154 on Day 29
  Interventions: Biological: ARCT-154
- Study Group 6, Adult Participants Previously Vaccinated randomized to receive ARCT-165 (Experimental): Participants will receive one dose of ARCT-165 on Day 1
  Interventions: Biological: ARCT-165
- Study Group 7, Adult Participants Previously Vaccinated randomized to receive ARCT-154 (Experimental): Participants will receive one dose of ARCT-154 on Day 1
  Interventions: Biological: ARCT-154
- Study Group 8, Adult Participants Previously Vaccinated randomized to receive ARCT-021 (Experimental): Participants will receive one dose of ARCT-021 on Day 1
  Interventions: Biological: ARCT-021

INTERVENTIONS:
Biological: ARCT-165 — Dose 3
  Arms: Study Group 1, Adult Participants Seronegative, Not Previously Vaccinated randomized to ARCT-165; Study Group 6, Adult Participants Previously Vaccinated randomized to receive ARCT-165
Biological: ARCT-154 — Dose 2
  Arms: Study Group 2, Adult Participants Seronegative, Not Previously Vaccinated randomized to ARCT-154; Study Group 5, Adult Participants Seropositive, Not Previously Vaccinated randomized to ARCT-154; Study Group 7, Adult Participants Previously Vaccinated randomized to receive ARCT-154
Biological: ARCT-021 — Dose 1
  Arms: Study Group 3, Adult Participants Seronegative, Not Previously Vaccinated to receive ARCT-021; Study Group 4, Adult Participants Seropositive, Not Previously Vaccinated to receive ARCT-021; Study Group 8, Adult Participants Previously Vaccinated randomized to receive ARCT-021

SUMMARY:
This is a Phase 1/2, randomized, observer-blind study in healthy adults. The study will evaluate the safety, reactogenicity, and immunogenicity of 3 SARS-CoV-2 self-amplifying RNA vaccine candidates against COVID-19 in adults previously vaccinated and not previously vaccinated against SARS-CoV-2.

DETAILED DESCRIPTION:
The study will initially enroll approximately 72 adult participants into 2 cohorts (A and B). Cohort A is further sub-divided into two sub-cohorts which include 12 participants who are seronegative, not previously vaccinated at screening (Sub-cohort A1) and 24 participants who are seropositive, not previously vaccinated at screening (Sub-cohort A2).

Within the first cohort (Cohort A), Sub-cohort A1 will include a total of 12 adult participants ≥21 to ≤65 years of age who have not been previously vaccinated with a SARS-CoV-2 vaccine. Sub-cohort A2 will include a total of 24 adult participants ≥21 to ≤65 years of age who have not been previously vaccinated with a SARS-CoV-2 vaccine. Study vaccines will be given as 2 doses separated by 28 days.

The second cohort (Cohort B) will include a total of 36 adult participants ≥21 to ≤65 years of age who have been previously vaccinated (5 months or longer prior to study enrollment) with SARS-CoV-2 vaccine. Study vaccines will be given as single doses.

Additional cohorts may increase the age range of participants up to 80 years of age.

ELIGIBILITY:
Inclusion Criteria:

Individuals who:

1. Are able to provide consent
2. Agree to comply with all study visits and procedures
3. Are willing and able to adhere to study restrictions
4. Are sexually active and willing to adhere to contraceptive requirements
5. Are male, female, or transgender ≥21 to ≤80 years of age
6. For the previously vaccinated groups only, received 2 doses of SARS-CoV-2 vaccine 5 months or longer prior to study enrollment

Exclusion Criteria:

Individuals who:

1. For the unvaccinated groups only, previously received any investigational or authorized MERS-CoV, SARS-CoV, and SARS-CoV-2 vaccines (including ARCT-021)
2. For the previously vaccinated groups only, previously received BNT162b2 but have not received 2 doses within at least 5 months prior to study enrollment
3. Are planning to receive other COVID-19 vaccines during the study period
4. Recently received other vaccines
5. Have a fever or are feeling sick close to the time of the first study vaccination
6. Have a known history of COVID-19 disease or asymptomatic SARS-CoV-2 infection
7. Are pregnant or breastfeeding
8. Have had a severe reaction to previous vaccines
9. Have a severe or uncontrolled disease(s) that may interfere with the interpretation of the study
10. Have some respiratory diseases
11. Have some significant heart diseases
12. Have some neurological conditions
13. Have sickle cell disease or some other blood disorders
14. Have had a major surgery within the past 6 months
15. Have a history of chronic liver disease
16. Have a history of autoimmune disease or immunodeficiency
17. Have received allergy injections, interferon, immunomodulators, cytotoxic drugs or other similar toxic drugs.
18. Have received blood products
19. Have a positive test for hepatitis B or C or human immunodeficiency virus
20. Have uncontrolled hypertension
21. Have had cancer except for cancers that were treated and that have low risk of returning
22. Are obese
23. Are Investigator site staff members, employees of Arcturus or the contract research organization (CRO) directly involved in the conduct of the study, or site staff members otherwise supervised by the Investigator or immediate family members of any of the previously mentioned individuals

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Arcturus Therapeutics
Locations (4):
- United States (2):
  - Arcturus Investigational Site 202, Wichita, Kansas
  - Arcturus Investigational Site 201, Kansas City, Missouri
- Arcturus Investigational Site 101, Singapore, Singapore
- Arcturus Investigational Site 301, Diepkloof, Soweto, South Africa

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be made available to study investigators at this time.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A1: ARCT-021: Participants ≥21 to ≤65 years of age who had not been previously vaccinated with a SARS-CoV-2 vaccine and were seronegative at screening were randomized to receive two doses of ARCT-021 on Days 1 and 29. ARCT-021 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Ancestral strain.
- Cohort A1: ARCT-165: Participants ≥21 to ≤65 years of age who had not been previously vaccinated with a SARS-CoV-2 vaccine and were seronegative at screening were randomized to receive two doses of ARCT-165 on Days 1 and 29. ARCT-165 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Beta variant.
- Cohort A1: ARCT-154: Participants ≥21 to ≤65 years of age who had not been previously vaccinated with a SARS-CoV-2 vaccine and were seronegative at screening were randomized to receive two doses of ARCT-154 on Days 1 and 29. ARCT-154 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Ancestral strain including the D614G mutation.
- Cohort A2: ARCT-021: Participants ≥21 to ≤65 years of age who had not been previously vaccinated with a SARS-CoV-2 vaccine and were seropositive at screening were randomized to receive two doses of ARCT-021 on Days 1 and 29. ARCT-021 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Ancestral strain.
- Cohort A2: ARCT-154: Participants ≥21 to ≤65 years of age who had not been previously vaccinated with a SARS-CoV-2 vaccine and were seropositive at screening were randomized to receive two doses of ARCT-154 on Days 1 and 29. ARCT-154 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Ancestral strain including the D614G mutation.
- Cohort B: ARCT-021: Participants ≥21 to ≤65 years of age who had been previously vaccinated (5 months or longer prior to study enrollment) with the BNT162b2 (Comirnaty) SARS-CoV-2 vaccine were randomized to receive a single dose of ARCT-021 on Day 1. ARCT-021 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Ancestral strain.
- Cohort B: ARCT-165: Participants ≥21 to ≤65 years of age who had been previously vaccinated (5 months or longer prior to study enrollment) with the BNT162b2 (Comirnaty) SARS-CoV-2 vaccine were randomized to receive a single dose of ARCT-165 on Day 1. ARCT-165 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Beta variant.
- Cohort B: ARCT-154: Participants ≥21 to ≤65 years of age who had been previously vaccinated (5 months or longer prior to study enrollment) with the BNT162b2 (Comirnaty) SARS-CoV-2 vaccine were randomized to receive a single dose of ARCT-154 on Day 1. ARCT-154 is a monovalent vaccine encoding for SARS-CoV-2 S glycoprotein of the Ancestral strain including the D614G mutation.
Period: Overall Study
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Started | 4 | 4 | 4 | 6 | 18 | 12 | 12 | 12
Received at Least 1 Dose of Study Drug | 4 | 4 | 4 | 6 | 18 | 12 | 12 | 12
Completed | 4 | 2 | 4 | 5 | 17 | 9 | 12 | 12
Not Completed | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Measured in the Safety Set (SS): The SS included all randomized participants who received at least one dose of the study vaccine. Assignment of participants to study vaccine group was based on the study vaccine actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 18 | 12 | 12 | 12 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (17) | 34 (10) | 50 (17) | 33 (9) | 31 (8) | 44 (16) | 50 (13) | 44 (13) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 4 | 10 | 9 | 6 | 7 | 42
  Male | 1 | 3 | 2 | 2 | 8 | 3 | 6 | 5 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 4 | 4 | 6 | 17 | 10 | 12 | 12 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 0 | 0 | 2 | 2 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 5 | 16 | 1 | 2 | 0 | 27
  White | 2 | 0 | 1 | 1 | 2 | 9 | 8 | 10 | 33
  More than one race | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Local or Systemic Adverse Events (AEs)
Description: Solicited local AEs were defined as injection site erythema, injection site pain, injection site induration, and injection site tenderness. Solicited systemic AEs were defined as arthralgia, chills, diarrhea, dizziness, fatigue, fever (categorized by measured body temperature), headache, myalgia, nausea and vomiting. Data are reported for the number of participants with solicited local and solicited systemic AEs. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 8 (7 days after first vaccine administration for Cohorts A1, A2 and B), and up to Day 36 (7 days after second vaccine administration for Cohorts A1 and A2)
Population: Measured in the SS: The SS included all randomized participants who received at least one dose of the study vaccine. Assignment of participants to study vaccine group was based on the study vaccine actually received. Number analyzed for Cohort B arms for AEs after Dose 2 = 0 as participants in this Cohort received only a single dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 18 | 12 | 12 | 12
Participants
  Any Solicited Local AE After Dose 1 | 3 | 4 | 3 | 5 | 10 | 12 | 10 | 10
  Any Solicited Local AE After Dose 2: number analyzed (Participants) | 4 | 4 | 4 | 6 | 18 | 0 | 0 | 0
  Any Solicited Local AE After Dose 2 | 2 | 2 | 4 | 6 | 10 |  |  |
  Any Solicited Systemic AE After Dose 1 | 3 | 3 | 1 | 5 | 9 | 12 | 9 | 11
  Any Solicited Systemic AE After Dose 2: number analyzed (Participants) | 4 | 4 | 4 | 6 | 18 | 0 | 0 | 0
  Any Solicited Systemic AE After Dose 2 | 2 | 2 | 3 | 5 | 10 |  |  |

2. Primary Outcome: Number of Participants Reporting Unsolicited AEs
Description: Unsolicited AEs were defined as any spontaneously reported or discovered AE. Data are reported for the number of participants with unsolicited AEs. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 29 (28 days after vaccine administration for Cohort B), and up to Day 57 (up to 28 days after each vaccine administration for Cohorts A1 and A2)
Population: Measured in the SS: The SS included all randomized participants who received at least one dose of the study vaccine. Assignment of participants to study vaccine group was based on the study vaccine actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 18 | 12 | 12 | 12
Participants | 3 | 3 | 2 | 4 | 15 | 9 | 9 | 10

3. Primary Outcome: Number of Participants Reporting Medically Attended Adverse Events (MAAEs), AEs Leading to Discontinuation From Study Vaccine/Study Withdrawal, or Serious Adverse Events (SAEs)
Description: An MAAE was an AE that led to an unscheduled visit (including a telemedicine visit) with a health care provider (HCP) (e.g., nurse, nurse practitioner, physician's assistant, physician), including visits to a study site for unscheduled assessments (e.g., rash assessment, abnormal laboratory follow up, coronavirus disease 2019 [COVID-19]) and visits to HCPs external to the study site (e.g., urgent care, primary care physician). An SAE was defined as any event that resulted in death, was immediately life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Through Final Visit (365 days after last study vaccine dose); up to a maximum of approximately 394 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 18 | 12 | 12 | 12
Participants
  Any MAAEs | 0 | 1 | 0 | 1 | 3 | 2 | 1 | 0
  Any AEs Leading to Discontinuation from Study Vaccine/Study Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAEs | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

4. Primary Outcome: Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) Serum Neutralizing Antibody Levels, Expressed as Geometric Mean Concentration (GMC)
Description: Blood samples were collected to assess participants' immune response. GMC data are reported for the pseudoviral D614G variant. Data are reported in international units per milliliter (IU/mL).
Time Frame: Baseline, Days 29, 57, 209, Final Visit (approx. Day 394) for Cohorts A1 and A2; Baseline, Days 15, 29, 91, 181, 271 and Final Visit (approx. Day 366) for Cohort B
Population: Immunogenicity Analysis Set, all eligible enrolled participants who received the specified number of doses of study vaccine to which they were assigned within the predefined window, had ≥1 valid/evaluable immunogenicity results after specified dose, had blood collection within an appropriate window after specified dose, and no other major protocol deviations. Overall number participants analyzed=participants evaluable for endpoint. Number analyzed=participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 3 | 4 | 6 | 18 | 12 | 12 | 12
IU/mL
  Pseudoviral D614G; Baseline | 8 [NA to NA] — Confidence interval data were non-estimable because baseline values were below the limit of quantification for all participants in the arm. | 8 [6 to 11] | 12 [4 to 33] | 421 [74 to 2383] | 455 [202 to 1028] | 87 [51 to 148] | 94 [29 to 301] | 114 [58 to 224]
  Pseudoviral D614G; Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Pseudoviral D614G; Day 15 |  |  |  |  |  | 1415 [927 to 2160] | 2019 [1179 to 3459] | 3474 [1577 to 7656]
  Pseudoviral D614G; Day 29: number analyzed (Participants) | 3 | 2 | 4 | 6 | 17 | 12 | 12 | 12
  Pseudoviral D614G; Day 29 | 36 [0 to 2715] | 9 [2 to 47] | 26 [6 to 107] | 1966 [592 to 6534] | 1949 [1026 to 3701] | 1741 [1001 to 3028] | 2202 [1170 to 4145] | 4200 [2274 to 7757]
  Pseudoviral D614G; Day 57: number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Pseudoviral D614G; Day 57 | 42 [2 to 998] | 87 [0 to 1334270362] | 70 [11 to 452] | 2038 [676 to 6143] | 3563 [2083 to 6096] |  |  |
  Pseudoviral D614G; Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 12
  Pseudoviral D614G; Day 91 |  |  |  |  |  | 1796 [1067 to 3024] | 1697 [840 to 3429] | 3427 [2113 to 5558]
  Pseudoviral D614G; Day 181: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 9
  Pseudoviral D614G; Day 181 |  |  |  |  |  | 1072 [450 to 2551] | 1534 [552 to 4260] | 3041 [1334 to 6932]
  Pseudoviral D614G; Day 209: number analyzed (Participants) | 4 | 0 | 3 | 4 | 16 | 0 | 0 | 0
  Pseudoviral D614G; Day 209 | 90 [2 to 3976] |  | 19 [4 to 85] | 1340 [100 to 17882] | 1402 [819 to 2402] |  |  |
  Pseudoviral D614G; Day 271: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 9
  Pseudoviral D614G; Day 271 |  |  |  |  |  | 611 [246 to 1518] | 2158 [1198 to 3888] | 1965 [789 to 4893]
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 7
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366) |  |  |  |  |  | 564 [232 to 1370] | 1924 [374 to 9900] | 2463 [870 to 6976]
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 2 | 3 | 11 | 0 | 0 | 0
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394) | 60 [2 to 2088] |  | 14 [0 to 3129] | 1000 [10 to 100036] | 1324 [671 to 2609] |  |  |

5. Primary Outcome: SARS-CoV-2 Serum Neutralizing Antibody Levels, Expressed as GMC
Description: Blood samples were collected to assess participants' immune response. GMC data are reported for the pseudoviral B.1.351 (beta) variant. Data are reported in arbitrary units per milliliter (AU/mL).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 3 | 4 | 6 | 18 | 12 | 12 | 12
AU/mL
  Pseudoviral B.1.351 (Beta); Baseline | 14 [NA to NA] — Confidence interval data were non-estimable because baseline values were below the limit of quantification for all participants in the arm. | 14 [NA to NA] — Confidence interval data were non-estimable because baseline values were below the limit of quantification for all participants in the arm. | 14 [13 to 15] | 402 [92 to 1761] | 442 [187 to 1042] | 38 [21 to 70] | 44 [15 to 130] | 60 [31 to 117]
  Pseudoviral B.1.351 (Beta); Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Pseudoviral B.1.351 (Beta); Day 15 |  |  |  |  |  | 554 [370 to 829] | 1479 [824 to 2652] | 1692 [905 to 3162]
  Pseudoviral B.1.351 (Beta); Day 29: number analyzed (Participants) | 3 | 2 | 4 | 6 | 17 | 12 | 12 | 12
  Pseudoviral B.1.351 (Beta); Day 29 | 17 [7 to 45] | 32 [0 to 1385422] | 17 [12 to 24] | 1926 [788 to 4710] | 1273 [615 to 2634] | 664 [447 to 986] | 1608 [940 to 2749] | 1768 [1061 to 2948]
  Pseudoviral B.1.351 (Beta); Day 57: number analyzed (Participants) | 4 | 2 | 3 | 6 | 15 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Day 57 | 21 [6 to 75] | 452 [0 to 1024516559] | 27 [10 to 71] | 2292 [991 to 5300] | 3237 [2123 to 4936] |  |  |
  Pseudoviral B.1.351 (Beta); Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 12
  Pseudoviral B.1.351 (Beta); Day 91 |  |  |  |  |  | 560 [326 to 960] | 1079 [559 to 2083] | 1376 [838 to 2260]
  Pseudoviral B.1.351 (Beta); Day 181: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 9
  Pseudoviral B.1.351 (Beta); Day 181 |  |  |  |  |  | 400 [142 to 1126] | 708 [219 to 2293] | 1202 [512 to 2819]
  Pseudoviral B.1.351 (Beta); Day 209: number analyzed (Participants) | 4 | 0 | 2 | 4 | 16 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Day 209 | 97 [3 to 3668] |  | 14 [13 to 16] | 1372 [185 to 10163] | 1438 [780 to 2652] |  |  |
  Pseudoviral B.1.351 (Beta); Day 271: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 9
  Pseudoviral B.1.351 (Beta); Day 271 |  |  |  |  |  | 175 [30 to 1036] | 829 [252 to 2724] | 1129 [446 to 2858]
  Pseudoviral B.1.351 (Beta); Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 8
  Pseudoviral B.1.351 (Beta); Final Visit Cohort B (approx. Day 366) |  |  |  |  |  | 213 [60 to 763] | 1532 [389 to 6036] | 1578 [604 to 4122]
  Pseudoviral B.1.351 (Beta); Final Visit Cohort A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 4 | 3 | 11 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Final Visit Cohort A1 and A2 (approx. Day 394) | 61 [3 to 1082] |  | 14 [NA to NA] — Confidence interval data were non-estimable because values were below the limit of quantification for all participants in the arm. | 1502 [45 to 50296] | 847 [467 to 1535] |  |  |

6. Primary Outcome: SARS-CoV-2 Serum Neutralizing Antibody Levels, Expressed as Geometric Mean Fold Rise (GMFR)
Description: Blood samples were collected to assess participants' immune response. GMFR data are reported for the pseudoviral D614G variant.
Time Frame: Days 29, 57, 209, Final Visit (approx. Day 394) for Cohorts A1 and A2, and Days 15, 29, 91, 181, 271 and Final Visit (approx. Day 366) for Cohort B
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 2 | 4 | 6 | 17 | 12 | 12 | 12
ratio
  Pseudoviral D614G; Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Pseudoviral D614G; Day 15 |  |  |  |  |  | 16 [9 to 30] | 22 [9 to 50] | 28 [11 to 67]
  Pseudoviral D614G; Day 29: number analyzed (Participants) | 3 | 2 | 4 | 6 | 17 | 12 | 12 | 12
  Pseudoviral D614G; Day 29 | 4.6 [0.1 to 346.2] | 1.0 [0.6 to 1.7] | 2.2 [0.4 to 12.2] | 4.7 [1.4 to 15.9] | 4.4 [2.7 to 7] | 20 [10 to 41] | 24 [10 to 54] | 37 [17 to 77]
  Pseudoviral D614G; Day 57: number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Pseudoviral D614G; Day 57 | 5.4 [0.2 to 127.2] | 10.1 [0 to 48765966.9] | 5.9 [0.5 to 65] | 4.8 [1.2 to 19.0] | 6.2 [3.8 to 10] |  |  |
  Pseudoviral D614G; Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 12
  Pseudoviral D614G; Day 91 |  |  |  |  |  | 20 [10 to 41] | 17 [8 to 36] | 30 [19 to 47]
  Pseudoviral D614G; Day 181: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 9
  Pseudoviral D614G; Day 181 |  |  |  |  |  | 11 [4 to 30] | 12 [3 to 45] | 31 [14 to 70]
  Pseudoviral D614G; Day 209: number analyzed (Participants) | 4 | 0 | 3 | 4 | 16 | 0 | 0 | 0
  Pseudoviral D614G; Day 209 | 11.4 [0.3 to 506.9] |  | 1.4 [0.1 to 14.7] | 3.2 [0.7 to 14.2] | 2.7 [1.8 to 4.1] |  |  |
  Pseudoviral D614G; Day 271: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 9
  Pseudoviral D614G; Day 271 |  |  |  |  |  | 5 [1 to 19] | 13 [2 to 71] | 20 [10 to 43]
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 7
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366) |  |  |  |  |  | 6 [1 to 27] | 27 [5 to 147] | 25 [7 to 88]
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 2 | 3 | 11 | 0 | 0 | 0
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394) | 7.7 [0.2 to 266.2] |  | 0.8 [0 to 329524.9] | 2.7 [0.2 to 42.6] | 1.9 [1.1 to 3.3] |  |  |

7. Primary Outcome: SARS-CoV-2 Serum Neutralizing Antibody Levels, Expressed as GMFR
Description: Blood samples were collected to assess participants' immune response. GMFR data are reported for the pseudoviral B.1.351 (beta) variant.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 2 | 4 | 6 | 17 | 12 | 12 | 12
ratio
  Pseudoviral B.1.351 (Beta); Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Pseudoviral B.1.351 (Beta); Day 15 |  |  |  |  |  | 14 [8 to 26] | 34 [16 to 72] | 25 [12 to 51]
  Pseudoviral B.1.351 (Beta); Day 29: number analyzed (Participants) | 3 | 2 | 4 | 6 | 17 | 12 | 12 | 12
  Pseudoviral B.1.351 (Beta); Day 29 | 1.2 [0.5 to 3.2] | 2.3 [0 to 98958.7] | 1.2 [0.8 to 1.7] | 4.8 [1.6 to 14.0] | 3.2 [1.3 to 7.5] | 17 [10 to 31] | 37 [17 to 77] | 29 [16 to 54]
  Pseudoviral B.1.351 (Beta); Day 57: number analyzed (Participants) | 4 | 2 | 3 | 6 | 15 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Day 57 | 1.5 [0.4 to 5.4] | 32.3 [0 to 73179754.2] | 1.9 [0.7 to 4.9] | 5.7 [1.4 to 22.7] | 5.6 [3.3 to 9.7] |  |  |
  Pseudoviral B.1.351 (Beta); Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 12
  Pseudoviral B.1.351 (Beta); Day 91 |  |  |  |  |  | 14 [7 to 27] | 23 [10 to 51] | 23 [15 to 35]
  Pseudoviral B.1.351 (Beta); Day 181: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 9
  Pseudoviral B.1.351 (Beta); Day 181 |  |  |  |  |  | 10 [4 to 26] | 12 [1 to 98] | 24 [10 to 56]
  Pseudoviral B.1.351 (Beta); Day 209: number analyzed (Participants) | 4 | 0 | 2 | 4 | 16 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Day 209 | 6.9 [0.2 to 262.0] |  | 1.0 [NA to NA] — Confidence interval data were non-estimable because values were below the limit of quantification for all participants in the arm. | 2.8 [0.7 to 11.6] | 2.9 [1.8 to 4.6] |  |  |
  Pseudoviral B.1.351 (Beta); Day 271: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 9
  Pseudoviral B.1.351 (Beta); Day 271 |  |  |  |  |  | 4 [2 to 8] | 12 [2 to 71] | 23 [11 to 45]
  Pseudoviral B.1.351 (Beta); Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 8
  Pseudoviral B.1.351 (Beta); Final Visit Cohort B (approx. Day 366) |  |  |  |  |  | 5 [1 to 22] | 46 [5 to 409] | 31 [9 to 108]
  Pseudoviral B.1.351 (Beta); Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 4 | 3 | 11 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Final Visit Cohorts A1 and A2 (approx. Day 394) | 4.4 [0.2 to 77.3] |  | 1.0 [0.6 to 1.5] | 3.0 [0.2 to 42.9] | 1.7 [0.9 to 3.2] |  |  |

8. Primary Outcome: Number of Participants Achieving Greater Than or Equal to 4-fold Rise From Before Vaccination in SARS-CoV-2 Serum Neutralizing Antibody Levels (Pseudoviral D614G Variant)
Description: Blood samples were collected to assess participants' immune response. Data are reported for the pseudoviral D614G variant.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 2 | 4 | 6 | 17 | 12 | 12 | 12
Participants
  Pseudoviral D614G; Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Pseudoviral D614G; Day 15 |  |  |  |  |  | 11 | 11 | 10
  Pseudoviral D614G; Day 29: number analyzed (Participants) | 3 | 2 | 4 | 6 | 17 | 12 | 12 | 12
  Pseudoviral D614G; Day 29 | 1 | 0 | 2 | 3 | 10 | 11 | 11 | 11
  Pseudoviral D614G; Day 57: number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Pseudoviral D614G; Day 57 | 2 | 1 | 2 | 4 | 11 |  |  |
  Pseudoviral D614G; Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 12
  Pseudoviral D614G; Day 91 |  |  |  |  |  | 10 | 10 | 12
  Pseudoviral D614G; Day 181: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 9
  Pseudoviral D614G; Day 181 |  |  |  |  |  | 5 | 8 | 9
  Pseudoviral D614G; Day 209: number analyzed (Participants) | 4 | 0 | 3 | 4 | 16 | 0 | 0 | 0
  Pseudoviral D614G; Day 209 | 2 |  | 0 | 1 | 5 |  |  |
  Pseudoviral D614G; Day 271: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 9
  Pseudoviral D614G; Day 271 |  |  |  |  |  | 3 | 6 | 8
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 7
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366) |  |  |  |  |  | 3 | 5 | 6
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 2 | 3 | 11 | 0 | 0 | 0
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394) | 2 |  | 0 | 1 | 1 |  |  |

9. Primary Outcome: Number of Participants Achieving Greater Than or Equal to 4-fold Rise From Before Vaccination in SARS-CoV-2 Serum Neutralizing Antibody Levels (Pseudoviral B.1.351 [Beta] Variant)
Description: Blood samples were collected to assess participants' immune response. Data are reported for the pseudoviral B.1.351 (beta) variant.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 2 | 4 | 6 | 17 | 12 | 12 | 12
Participants
  Pseudoviral B.1.351 (Beta); Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Pseudoviral B.1.351 (Beta); Day 15 |  |  |  |  |  | 11 | 11 | 10
  Pseudoviral B.1.351 (Beta); Day 29: number analyzed (Participants) | 3 | 2 | 4 | 6 | 17 | 12 | 12 | 12
  Pseudoviral B.1.351 (Beta); Day 29 | 0 | 1 | 0 | 3 | 9 | 11 | 11 | 11
  Pseudoviral B.1.351 (Beta); Day 57: number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Day 57 | 1 | 2 | 1 | 3 | 9 |  |  |
  Pseudoviral B.1.351 (Beta); Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 12
  Pseudoviral B.1.351 (Beta); Day 91 |  |  |  |  |  | 9 | 10 | 12
  Pseudoviral B.1.351 (Beta); Day 181: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 9
  Pseudoviral B.1.351 (Beta); Day 181 |  |  |  |  |  | 4 | 8 | 8
  Pseudoviral B.1.351 (Beta); Day 209: number analyzed (Participants) | 4 | 0 | 3 | 4 | 16 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Day 209 | 2 |  | 0 | 1 | 5 |  |  |
  Pseudoviral B.1.351 (Beta); Day 271: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 9
  Pseudoviral B.1.351 (Beta); Day 271 |  |  |  |  |  | 2 | 5 | 9
  Pseudoviral B.1.351 (Beta); Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 8
  Pseudoviral B.1.351 (Beta); Final Visit Cohort B (approx. Day 366) |  |  |  |  |  | 3 | 4 | 7
  Pseudoviral B.1.351 (Beta); Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 2 | 3 | 11 | 0 | 0 | 0
  Pseudoviral B.1.351 (Beta); Final Visit Cohorts A1 and A2 (approx. Day 394) | 2 |  | 0 | 1 | 1 |  |  |

10. Primary Outcome: GMC Ratio (ARCT-165 vs ARCT-154 and ARCT-021 vs ARCT-154)
Description: Blood samples were collected to assess participants' immune response. Data are reported for the pseudoviral D614G Variant, B.1.351 Variant, B.1.617.2 Variant, BA.1 Variant for the GMC ratio of ARCT-165 vs ARCT-154 and ARCT-021 vs ARCT-154. Data are reported for the ARCT-165 and ARCT-021 arms (vs ARCT-154 values).
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A2: ARCT-021 | Cohort B: ARCT-021 | Cohort B: ARCT-165
Number analyzed (Participants) | 4 | 2 | 6 | 12 | 12
ratio
  Pseudoviral D614G; Day 15: number analyzed (Participants) | 0 | 0 | 0 | 12 | 12
  Pseudoviral D614G; Day 15 |  |  |  | 0.41 [0.179 to 0.924] | 0.58 [0.240 to 1.405]
  Pseudoviral D614G; Day 29: number analyzed (Participants) | 3 | 2 | 6 | 12 | 12
  Pseudoviral D614G; Day 29 | 1.38 [0.108 to 17.701] | 0.35 [0.054 to 2.225] | 1.01 [0.301 to 3.377] | 0.41 [0.190 to 0.903] | 0.52 [0.229 to 1.203]
  Pseudoviral D614G; Day 57: number analyzed (Participants) | 4 | 2 | 6 | 0 | 0
  Pseudoviral D614G; Day 57 | 0.60 [0.035 to 10.082] | 1.23 [0.046 to 33.164] | 0.57 [0.210 to 1.559] |  |
  Pseudoviral D614G; Day 91: number analyzed (Participants) | 0 | 0 | 0 | 10 | 11
  Pseudoviral D614G; Day 91 |  |  |  | 0.52 [0.269 to 1.021] | 0.50 [0.225 to 1.089]
  Pseudoviral D614G; Day 181: number analyzed (Participants) | 0 | 0 | 0 | 6 | 9
  Pseudoviral D614G; Day 181 |  |  |  | 0.35 [0.115 to 1.082] | 0.50 [0.151 to 1.686]
  Pseudoviral D614G; Day 209: number analyzed (Participants) | 4 | 0 | 4 | 0 | 0
  Pseudoviral D614G; Day 209 | 4.65 [0.115 to 188.134] |  | 0.96 [0.251 to 3.629] |  |
  Pseudoviral D614G; Day 271: number analyzed (Participants) | 0 | 0 | 0 | 5 | 7
  Pseudoviral D614G; Day 271 |  |  |  | 0.31 [0.086 to 1.123] | 1.10 [0.377 to 3.199]
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 3 | 0 | 0
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394) | 4.20 [0.038 to 458.249] |  | 0.76 [0.139 to 4.106] |  |
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 5 | 5
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366) |  |  |  | 0.23 [0.064 to 0.825] | 0.78 [0.162 to 3.771]
  Pseudoviral B.1.351; Day 15: number analyzed (Participants) | 0 | 0 | 0 | 12 | 12
  Pseudoviral B.1.351; Day 15 |  |  |  | 0.33 [0.165 to 0.650] | 0.87 [0.392 to 1.951]
  Pseudoviral B.1.351; Day 29: number analyzed (Participants) | 3 | 2 | 6 | 12 | 12
  Pseudoviral B.1.351; Day 29 | 1.03 [0.575 to 1.846] | 1.92 [0.426 to 8.609] | 1.51 [0.418 to 5.476] | 0.38 [0.204 to 0.691] | 0.91 [0.452 to 1.827]
  Pseudoviral B.1.351; Day 57: number analyzed (Participants) | 4 | 2 | 6 | 0 | 0
  Pseudoviral B.1.351; Day 57 | 0.78 [0.227 to 2.712] | 16.96 [1.632 to 176.241] | 0.71 [0.325 to 1.545] |  |
  Pseudoviral B.1.351; Day 91: number analyzed (Participants) | 0 | 0 | 0 | 10 | 11
  Pseudoviral B.1.351; Day 91 |  |  |  | 0.41 [0.205 to 0.808] | 0.78 [0.365 to 1.684]
  Pseudoviral B.1.351; Day 181: number analyzed (Participants) | 0 | 0 | 0 | 6 | 9
  Pseudoviral B.1.351; Day 181 |  |  |  | 0.33 [0.099 to 1.117] | 0.59 [0.155 to 2.238]
  Pseudoviral B.1.351; Day 209: number analyzed (Participants) | 4 | 0 | 4 | 0 | 0
  Pseudoviral B.1.351; Day 209 | 6.77 [0.210 to 218.085] |  | 0.95 [0.242 to 3.759] |  |
  Pseudoviral B.1.351; Day 271: number analyzed (Participants) | 0 | 0 | 0 | 5 | 7
  Pseudoviral B.1.351; Day 271 |  |  |  | 0.16 [0.032 to 0.742] | 0.73 [0.192 to 2.813]
  Pseudoviral B.1.351; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 3 | 0 | 0
  Pseudoviral B.1.351; Final Visit Cohorts A1 and A2 (approx. Day 394) | 4.37 [0.102 to 187.648] |  | 1.77 [0.433 to 7.256] |  |
  Pseudoviral B.1.351; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 6 | 5
  Pseudoviral B.1.351; Final Visit Cohort B (approx. Day 366) |  |  |  | 0.14 [0.034 to 0.540] | 0.97 [0.234 to 4.022]
  Pseudoviral B.1.617.2; Day 15: number analyzed (Participants) | 0 | 0 | 0 | 12 | 12
  Pseudoviral B.1.617.2; Day 15 |  |  |  | 0.43 [0.208 to 0.900] | 0.69 [0.293 to 1.611]
  Pseudoviral B.1.617.2; Day 29: number analyzed (Participants) | 3 | 2 | 6 | 12 | 12
  Pseudoviral B.1.617.2; Day 29 | 2.45 [0.183 to 32.786] | 0.77 [0.268 to 2.241] | 1.17 [0.386 to 3.544] | 0.47 [0.231 to 0.947] | 0.66 [0.305 to 1.447]
  Pseudoviral B.1.617.2; Day 57: number analyzed (Participants) | 4 | 2 | 6 | 0 | 0
  Pseudoviral B.1.617.2; Day 57 | 1.78 [0.293 to 10.846] | 1.42 [0.552 to 3.644] | 0.92 [0.345 to 2.469] |  |
  Pseudoviral B.1.617.2; Day 91: number analyzed (Participants) | 0 | 0 | 0 | 10 | 11
  Pseudoviral B.1.617.2; Day 91 |  |  |  | 0.68 [0.266 to 1.740] | 0.61 [0.277 to 1.331]
  Pseudoviral B.1.617.2; Day 181: number analyzed (Participants) | 0 | 0 | 0 | 6 | 9
  Pseudoviral B.1.617.2; Day 181 |  |  |  | 0.46 [0.142 to 1.466] | 0.82 [0.274 to 2.465]
  Pseudoviral B.1.617.2; Day 209: number analyzed (Participants) | 4 | 0 | 4 | 0 | 0
  Pseudoviral B.1.617.2; Day 209 | 3.26 [0.388 to 27.333] |  | 0.59 [0.116 to 3.053] |  |
  Pseudoviral B.1.617.2; Day 271: number analyzed (Participants) | 0 | 0 | 0 | 5 | 7
  Pseudoviral B.1.617.2; Day 271 |  |  |  | 0.41 [0.114 to 1.465] | 1.30 [0.482 to 3.497]
  Pseudoviral B.1.617.2; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 3 | 0 | 0
  Pseudoviral B.1.617.2; Final Visit Cohorts A1 and A2 (approx. Day 394) | 2.18 [0.317 to 15.035] |  | 0.84 [0.179 to 3.905] |  |
  Pseudoviral B.1.617.2; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 6 | 5
  Pseudoviral B.1.617.2; Final Visit Cohort B (approx. Day 366) |  |  |  | 0.35 [0.095 to 1.282] | 1.30 [0.279 to 6.100]
  Pseudoviral BA.1 Variant; Day 15: number analyzed (Participants) | 0 | 0 | 0 | 12 | 12
  Pseudoviral BA.1 Variant; Day 15 |  |  |  | 0.34 [0.159 to 0.740] | 1.18 [0.501 to 2.799]
  Pseudoviral BA.1 Variant; Day 29: number analyzed (Participants) | 3 | 2 | 6 | 12 | 12
  Pseudoviral BA.1 Variant; Day 29 | 1.52 [0.677 to 3.427] | 1.05 [0.832 to 1.336] | 1.18 [0.369 to 3.760] | 0.36 [0.182 to 0.703] | 1.06 [0.485 to 2.310]
  Pseudoviral BA.1 Variant; Day 57: number analyzed (Participants) | 4 | 2 | 6 | 0 | 0
  Pseudoviral BA.1 Variant; Day 57 | 1.15 [0.612 to 2.153] | 9.73 [0.286 to 331.151] | 0.74 [0.287 to 1.913] |  |
  Pseudoviral BA.1 Variant; Day 91: number analyzed (Participants) | 0 | 0 | 0 | 10 | 11
  Pseudoviral BA.1 Variant; Day 91 |  |  |  | 0.35 [0.182 to 0.666] | 0.82 [0.361 to 1.856]
  Pseudoviral BA.1 Variant; Day 181: number analyzed (Participants) | 0 | 0 | 0 | 6 | 9
  Pseudoviral BA.1 Variant; Day 181 |  |  |  | 0.22 [0.047 to 1.032] | 0.82 [0.194 to 3.479]
  Pseudoviral BA.1 Variant; Day 209: number analyzed (Participants) | 4 | 0 | 4 | 0 | 0
  Pseudoviral BA.1 Variant; Day 209 | 8.15 [0.701 to 94.646] |  | 1.38 [0.260 to 7.365] |  |
  Pseudoviral BA.1 Variant; Day 271: number analyzed (Participants) | 0 | 0 | 0 | 5 | 7
  Pseudoviral BA.1 Variant; Day 271 |  |  |  | 0.20 [0.038 to 1.011] | 1.27 [0.369 to 4.347]
  Pseudoviral BA.1 Variant; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0 | 3 | 0 | 0
  Pseudoviral BA.1 Variant; Final Visit Cohorts A1 and A2 (approx. Day 394) | 3.69 [0.190 to 71.730] |  | 1.91 [0.223 to 16.385] |  |
  Pseudoviral BA.1 Variant; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 0 | 0 | 6 | 5
  Pseudoviral BA.1 Variant; Final Visit Cohort B (approx. Day 366) |  |  |  | 0.11 [0.020 to 0.562] | 0.87 [0.162 to 4.620]

11. Primary Outcome: GMC Ratio (ARCT-021 vs ARCT-165 Cohorts A1 and B)
Description: Blood samples were collected to assess participants' immune response. Data are reported for the pseudoviral D614G Variant, B.1.351 Variant, B.1.617.2 Variant, BA.1 Variant for the GMC ratio of ARCT-021 vs ARCT-165. Data are reported for the ARCT-021 arm (vs ARCT-165 values).
Time Frame: Days 29, 57, 209, Final Visit (approx. Day 394) for Cohort A1, and Days 15, 29, 91, 181, 271 and Final Visit (approx. Day 366) for Cohort B
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: ARCT-021 | Cohort B: ARCT-021
Number analyzed (Participants) | 4 | 12
ratio
  Pseudoviral D614G; Day 15: number analyzed (Participants) | 0 | 12
  Pseudoviral D614G; Day 15 |  | 0.70 [0.368 to 1.335]
  Pseudoviral D614G; Day 29: number analyzed (Participants) | 3 | 12
  Pseudoviral D614G; Day 29 | 4.00 [0.063 to 252.690] | 0.79 [0.358 to 1.746]
  Pseudoviral D614G; Day 57: number analyzed (Participants) | 4 | 0
  Pseudoviral D614G; Day 57 | 0.48 [0.004 to 53.354] |
  Pseudoviral D614G; Day 91: number analyzed (Participants) | 0 | 10
  Pseudoviral D614G; Day 91 |  | 1.06 [0.460 to 2.432]
  Pseudoviral D614G; Day 181: number analyzed (Participants) | 0 | 6
  Pseudoviral D614G; Day 181 |  | 0.70 [0.186 to 2.624]
  Pseudoviral D614G; Day 209: number analyzed (Participants) | 4 | 0
  Pseudoviral D614G; Day 209 | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral D614G; Day 271: number analyzed (Participants) | 0 | 5
  Pseudoviral D614G; Day 271 |  | 0.28 [0.117 to 0.684]
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0
  Pseudoviral D614G; Final Visit Cohorts A1 and A2 (approx. Day 394) | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 5
  Pseudoviral D614G; Final Visit Cohort B (approx. Day 366) |  | 0.29 [0.062 to 1.377]
  Pseudoviral B.1.351; Day 15: number analyzed (Participants) | 0 | 12
  Pseudoviral B.1.351; Day 15 |  | 0.37 [0.192 to 0.731]
  Pseudoviral B.1.351; Day 29: number analyzed (Participants) | 3 | 12
  Pseudoviral B.1.351; Day 29 | 0.54 [0.061 to 4.779] | 0.41 [0.221 to 0.774]
  Pseudoviral B.1.351; Day 57: number analyzed (Participants) | 4 | 0
  Pseudoviral B.1.351; Day 57 | 0.05 [0.004 to 0.609] |
  Pseudoviral B.1.351; Day 91: number analyzed (Participants) | 0 | 10
  Pseudoviral B.1.351; Day 91 |  | 0.52 [0.232 to 1.160]
  Pseudoviral B.1.351; Day 181: number analyzed (Participants) | 0 | 6
  Pseudoviral B.1.351; Day 181 |  | 0.56 [0.122 to 2.616]
  Pseudoviral B.1.351; Day 209: number analyzed (Participants) | 4 | 0
  Pseudoviral B.1.351; Day 209 | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral B.1.351; Day 271: number analyzed (Participants) | 0 | 5
  Pseudoviral B.1.351; Day 271 |  | 0.21 [0.037 to 1.223]
  Pseudoviral B.1.351; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0
  Pseudoviral B.1.351; Final Visit Cohorts A1 and A2 (approx. Day 394) | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral B.1.351; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 6
  Pseudoviral B.1.351; Final Visit Cohort B (approx. Day 366) |  | 0.14 [0.028 to 0.688]
  Pseudoviral B.1.617.2; Day 15: number analyzed (Participants) | 0 | 12
  Pseudoviral B.1.617.2; Day 15 |  | 0.63 [0.328 to 1.210]
  Pseudoviral B.1.617.2; Day 29: number analyzed (Participants) | 3 | 12
  Pseudoviral B.1.617.2; Day 29 | 3.16 [0.028 to 357.696] | 0.70 [0.365 to 1.357]
  Pseudoviral B.1.617.2; Day 57: number analyzed (Participants) | 4 | 0
  Pseudoviral B.1.617.2; Day 57 | 1.26 [0.053 to 29.735] |
  Pseudoviral B.1.617.2; Day 91: number analyzed (Participants) | 0 | 10
  Pseudoviral B.1.617.2; Day 91 |  | 0.68 [0.266 to 1.740]
  Pseudoviral B.1.617.2; Day 181: number analyzed (Participants) | 0 | 6
  Pseudoviral B.1.617.2; Day 181 |  | 0.56 [0.159 to 1.948]
  Pseudoviral B.1.617.2; Day 209: number analyzed (Participants) | 4 | 0
  Pseudoviral B.1.617.2; Day 209 | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral B.1.617.2; Day 271: number analyzed (Participants) | 0 | 5
  Pseudoviral B.1.617.2; Day 271 |  | 0.31 [0.109 to 0.904]
  Pseudoviral B.1.617.2; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0
  Pseudoviral B.1.617.2; Final Visit Cohorts A1 and A2 (approx. Day 394) | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral B.1.617.2; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 6
  Pseudoviral B.1.617.2; Final Visit Cohort B (approx. Day 366) |  | 0.27 [0.065 to 1.097]
  Pseudoviral BA.1 Variant; Day 15: number analyzed (Participants) | 0 | 12
  Pseudoviral BA.1 Variant; Day 15 |  | 0.29 [0.156 to 0.537]
  Pseudoviral BA.1 Variant; Day 29: number analyzed (Participants) | 3 | 12
  Pseudoviral BA.1 Variant; Day 29 | 1.45 [0.304 to 6.868] | 0.34 [0.174 to 0.654]
  Pseudoviral BA.1 Variant; Day 57: number analyzed (Participants) | 4 | 0
  Pseudoviral BA.1 Variant; Day 57 | 0.12 [0.003 to 4.660] |
  Pseudoviral BA.1 Variant; Day 91: number analyzed (Participants) | 0 | 10
  Pseudoviral BA.1 Variant; Day 91 |  | 0.43 [0.182 to 0.996]
  Pseudoviral BA.1 Variant; Day 181: number analyzed (Participants) | 0 | 6
  Pseudoviral BA.1 Variant; Day 181 |  | 0.27 [0.059 to 1.217]
  Pseudoviral BA.1 Variant; Day 209: number analyzed (Participants) | 4 | 0
  Pseudoviral BA.1 Variant; Day 209 | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral BA.1 Variant; Day 271: number analyzed (Participants) | 0 | 5
  Pseudoviral BA.1 Variant; Day 271 |  | 0.15 [0.042 to 0.570]
  Pseudoviral BA.1 Variant; Final Visit Cohorts A1 and A2 (approx. Day 394): number analyzed (Participants) | 4 | 0
  Pseudoviral BA.1 Variant; Final Visit Cohorts A1 and A2 (approx. Day 394) | NA [NA to NA] — Data were non-estimable because values were below the limit of quantification for all participants in the arm. |
  Pseudoviral BA.1 Variant; Final Visit Cohort B (approx. Day 366): number analyzed (Participants) | 0 | 6
  Pseudoviral BA.1 Variant; Final Visit Cohort B (approx. Day 366) |  | 0.12 [0.024 to 0.622]

12. Primary Outcome: SARS-CoV-2 Full-length Spike and Receptor-binding Domain (RBD) Binding Antibody Levels, Expressed as GMCs
Description: Spike binding antibody levels expressed as GMCs are reported for ancestral, D614G, and B.1.351 variants and RBD binding antibodies for ancestral strain.
Time Frame: Baseline and Day 57 for Cohorts A1 and A2, Baseline and Day 15 for Cohort B
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 3 | 4 | 6 | 18 | 12 | 12 | 12
AU/mL
  Baseline; RBD (Ancestral) | 0.0 [0.0 to 0.0] | 0.1 [0.0 to 1.2] | 0.1 [0.0 to 0.7] | 34 [9 to 124] | 29 [14 to 60] | 9 [6 to 14] | 9 [4 to 21] | 10 [6 to 16]
  Baseline; Spike (Ancestral) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.4] | 0.3 [0.0 to 1.7] | 44 [13 to 156] | 49 [27 to 90] | 18 [12 to 27] | 17 [8 to 39] | 19 [11 to 33]
  Baseline; Spike (D614G) | 0.0 [0.0 to 0.2] | 0.1 [0.0 to 0.9] | 0.2 [0.0 to 1.7] | 47 [14 to 161] | 52 [29 to 95] | 19 [13 to 27] | 18 [8 to 40] | 20 [11 to 35]
  Baseline; Spike (B.1.351) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.5] | 0.2 [0.0 to 1.6] | 30 [11 to 77] | 32 [19 to 56] | 8 [6 to 12] | 8 [4 to 17] | 9 [5 to 16]
  Day 57; RBD (Ancestral): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; RBD (Ancestral) | 3.4 [0.1 to 133.7] | 34.5 [0.0 to 13491400] | 8.2 [1.2 to 54.5] | 138 [49 to 386] | 186 [128 to 270] |  |  |
  Day 57; Spike (Ancestral): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (Ancestral) | 10.6 [0.4 to 285.1] | 52.4 [0.0 to 3217076.2] | 19.1 [3.3 to 108.8] | 181 [65 to 504] | 265 [196 to 358] |  |  |
  Day 57; Spike (D614G): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (D614G) | 10.7 [0.4 to 276.8] | 55.8 [0.0 to 1948962.5] | 19.8 [3.6 to 110.4] | 187 [69 to 511] | 277 [205 to 375] |  |  |
  Day 57; Spike (B.1.351): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (B.1.351) | 5.0 [0.2 to 147.4] | 61.1 [0.0 to 7370140.4] | 5.8 [0.6 to 58.4] | 119 [51 to 278] | 147 [112 to 193] |  |  |
  Day 15; RBD (Ancestral): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; RBD (Ancestral) |  |  |  |  |  | 91 [57 to 146] | 171 [115 to 254] | 221 [118 to 415]
  Day 15; Spike (Ancestral): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (Ancestral) |  |  |  |  |  | 138 [89 to 215] | 231 [150 to 355] | 290 [164 to 514]
  Day 15; Spike (D614G): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (D614G) |  |  |  |  |  | 142 [92 to 217] | 235 [154 to 359] | 296 [166 to 529]
  Day 15; Spike (B.1.351): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (B.1.351) |  |  |  |  |  | 57 [40 to 82] | 117 [79 to 172] | 123 [71 to 212]

13. Primary Outcome: Changes in SARS-CoV-2 Full-length Spike and RBD Binding Antibody Levels, Expressed as GMFRs
Description: Spike binding antibody levels expressed as GMFRs are reported for ancestral, D614G, and B.1.351 variants and RBD binding antibody levels expressed as GMFR for ancestral strain.
Time Frame: Day 57 for Cohorts A1 and A2, Day 15 for Cohort B
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 12 | 12 | 11
ratio
  Day 57; RBD (Ancestral): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; RBD (Ancestral) | 129 [6 to 2894] | 286 [0 to 46860600000] | 110 [8 to 1560] | 4.1 [1.4 to 12.3] | 4.9 [3.0 to 8.0] |  |  |
  Day 57; Spike (Ancestral): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (Ancestral) | 231 [10 to 5236] | 807 [0 to 184116000000] | 76 [5 to 1279] | 4.1 [1.6 to 10.8] | 4.2 [2.8 to 6.3] |  |  |
  Day 57; Spike (D614G): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (D614G) | 237 [10 to 5730] | 667 [0 to 2176320000000] | 84 [5 to 1404] | 4.0 [1.5 to 10.4] | 4.1 [2.8 to 6.1] |  |  |
  Day 57; Spike (B.1.351): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (B.1.351) | 136 [5 to 4083] | 1076 [0 to 12500400000000] | 32 [3 to 361] | 4.0 [1.6 to 10.2] | 3.6 [2.4 to 5.4] |  |  |
  Day 15; RBD (Ancestral): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; RBD (Ancestral) |  |  |  |  |  | 10 [6 to 16] | 19 [10 to 38] | 21 [11 to 40]
  Day 15; Spike (Ancestral): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (Ancestral) |  |  |  |  |  | 8 [5 to 13] | 13 [7 to 25] | 14 [8 to 26]
  Day 15; Spike (D614G): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (D614G) |  |  |  |  |  | 8 [5 to 13] | 13 [7 to 25] | 14 [7 to 26]
  Day 15; Spike (B.1.351): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (B.1.351) |  |  |  |  |  | 7 [4 to 11] | 15 [8 to 27] | 13 [7 to 22]

14. Primary Outcome: Number of Participants Achieving Greater Than or Equal to 4-fold Rise From Before Vaccination in SARS-CoV-2 Full-length Spike and RBD Binding Antibody Levels
Description: Data are reported for ancestral, D614G, and B.1.351 variants for Spike binding antibodies and ancestral for RBD binding antibodies.
Time Frame: Day 57 for Cohorts A1 and A2, Day 15 for Cohort B
Population: Immunogenicity Analysis Set, all eligible enrolled participants who received the specified number of doses of study vaccine to which they were assigned within the predefined window, had ≥1 valid/evaluable immunogenicity results after specified dose, had blood collection within an appropriate window after specified dose, and no other major protocol deviations. Overall number participants analyzed =participants evaluable for endpoint. Number analyzed =participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
Number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 12 | 12 | 11
Participants
  Day 57; RBD (Ancestral): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; RBD (Ancestral) | 4 | 2 | 4 | 3 | 9 |  |  |
  Day 57; Spike (Ancestral): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (Ancestral) | 4 | 2 | 4 | 3 | 8 |  |  |
  Day 57; Spike (D614G): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (D614G) | 4 | 2 | 4 | 3 | 8 |  |  |
  Day 57; Spike (B.1.351): number analyzed (Participants) | 4 | 2 | 4 | 6 | 15 | 0 | 0 | 0
  Day 57; Spike (B.1.351) | 4 | 2 | 4 | 3 | 6 |  |  |
  Day 15; RBD (Ancestral): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; RBD (Ancestral) |  |  |  |  |  | 11 | 11 | 10
  Day 15; Spike (Ancestral): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (Ancestral) |  |  |  |  |  | 9 | 10 | 10
  Day 15; Spike (D614G): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (D614G) |  |  |  |  |  | 9 | 11 | 10
  Day 15; Spike (B.1.351): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11
  Day 15; Spike (B.1.351) |  |  |  |  |  | 9 | 11 | 10

ADVERSE EVENTS:
Time Frame: Through Final Visit (365 days after last study vaccine dose); up to a maximum of approximately 394 days
Description: Measured in the SS: The SS included all randomized participants who received at least one dose of the study vaccine. Assignment of participants to study vaccine group was based on the study vaccine actually received.
Arm/Group | Cohort A1: ARCT-021 | Cohort A1: ARCT-165 | Cohort A1: ARCT-154 | Cohort A2: ARCT-021 | Cohort A2: ARCT-154 | Cohort B: ARCT-021 | Cohort B: ARCT-165 | Cohort B: ARCT-154
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/6 | 0/18 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 1/6 | 0/18 | 1/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 2/4 | 4/6 | 15/18 | 9/12 | 9/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort A1: ARCT-021 (N=4) | Cohort A1: ARCT-165 (N=4) | Cohort A1: ARCT-154 (N=4) | Cohort A2: ARCT-021 (N=6) | Cohort A2: ARCT-154 (N=18) | Cohort B: ARCT-021 (N=12) | Cohort B: ARCT-165 (N=12) | Cohort B: ARCT-154 (N=12)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0/3 | 0/1 | 0/2 | 1/4 | 0/10 | 0/9 | 0/6 | 0/7 — N values for at risk have been adjusted as this is a sex-specific event.
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: ARCT-021 (N=4) | Cohort A1: ARCT-165 (N=4) | Cohort A1: ARCT-154 (N=4) | Cohort A2: ARCT-021 (N=6) | Cohort A2: ARCT-154 (N=18) | Cohort B: ARCT-021 (N=12) | Cohort B: ARCT-165 (N=12) | Cohort B: ARCT-154 (N=12)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 15 | 0 | 1 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 6 | 4 | 6 | 6
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericoronitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 2 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 5 | 1 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 2 | 2 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral lichen planus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05037097/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT05037097/SAP_001.pdf